CLINICAL TRIAL: NCT06654258
Title: Supporting Spiritual Wellbeing in Young Adults With Cancer Using a Digital Health Approach: A Feasibility Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Smartphone application being tested in this study was removed from commercial use
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00114969
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Young Adult Cancer
Keywords: spirituality; digital health; young adults; spiritual wellbeing; psychosocial wellbeing; young adult cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spiritual Self-Care App (Experimental): Smartphone app
  Interventions: Behavioral: Spiritual Self-Care Smartphone App

INTERVENTIONS:
Behavioral: Spiritual Self-Care Smartphone App — Participants will be asked to engage with a commercially available spiritual self-care smartphone app on a daily basis for 6 weeks. The content spans several domains, including meditation, prayer, affirmations, movement (i.e., stretching and yoga), and music. The user experience is highly personalized, allowing the user to select content that matches their current: mood or needs (e.g., anxiety, loneliness, stress, self-esteem, and sleep), time of day (e.g., recommendations for morning and evening practices), and/or availability (e.g., very brief "micro-interventions" lasting no more than 90 seconds or longer activities up to 30 minutes in duration). The content is delivered via a combination of audio and visual modalities on a personal smartphone that can be toggled on and off to adjust to surroundings.

SUMMARY:
The purpose of this research study is to collect information on how young adults (aged 18-39) receiving treatment for cancer use and rate the acceptability of a spiritual self-care smartphone app over a 6-week period. This study will test whether there may be any immediate or lasting benefits to spiritual or psychological wellbeing after using the app for 6-weeks. Collecting this information about the spiritual self-care app from young adults receiving treatment for cancer to better understand whether further testing of this smartphone app for supporting spiritual wellbeing during cancer treatment should be considered.

DETAILED DESCRIPTION:
On average, approximately 80,000 young adults (YAs) aged 18 to 39 are diagnosed with cancer each year in the USA, accounting for approximately 5% of all cancer diagnoses. YAs experience difficulties in dealing with the physical and psychological changes associated with cancer and its treatments, the management of acute and ongoing symptoms, and worrying about progression or recurrence. In addition, YAs are also engaging in normal developmental processes across various social, emotional, and financial domains. When diagnosed with cancer, these developmental processes are disrupted, resulting in elevated psychological and psychosocial distress. Although the reported quality and severity of these impacts are largely qualitative in nature, some reports indicate that YAs diagnosed with cancer are 57% more likely to develop depression and 29% more likely to develop anxiety than YAs without cancer and are more likely to have clinically significant levels of psychological distress compared to pediatric and older adults with cancer. To ensure the needs of this population are being met, it is important that supportive interventions for YAs with cancer are acceptable and age appropriate.

Spirituality refers to an individual's search for meaning in life and personal connectedness with the divine and transcendence beyond self, other individuals, and the environment and is recognized as an essential element of person-centered care. During developmental years, it is natural for YAs to explore spirituality to inform decisions, self-understanding, and meaning-making processes, and recent survey data from a nationally representative sample indicates that >50% of YAs report spirituality as important to them. Research has revealed that higher levels of spirituality predict better health-related quality of life in patients with cancer, even after accounting for physical and emotional wellbeing, and better patient reported mental health. However, there has been limited research exploring the unique spiritual perspectives of YAs resulting in insufficient guidance on how to best support them within this domain. Given the potential for spirituality to improve mental and physical health and to help reduce the psychosocial burden of a cancer diagnosis, research exploring spiritual self-care interventions in YAs with cancer is warranted.

Cancer patients report that they receive less spiritual care than desired from their healthcare providers. Research exploring barriers to delivering spiritual care at the bedside include time constraints, lack of confidence in effectiveness, and role uncertainty. When it comes to accessing spiritual care that is available, there are additional barriers for patients including: 1) requiring personal resources to access (e.g., transportation, time, insurance), or 2) limited options for remote, on-demand interventions despite preferences for them. Overall, there is a need and demand for accessible spiritual self-care for YAs, and addressing this gap could result in additional positive impacts on several aspects of physical and psychosocial wellbeing.

Digital health tools (e.g., smartphone apps) provide an opportunity to overcome barriers relevant to YAs with cancer including geographic mobility, time constraints, competing priorities, and limited psychosocial support providers. Furthermore, as 'digital natives', YAs are already high utilizers of technology, reducing the barrier of digital literacy in the uptake of such tools. Given the increasing focus on providing personalized, inclusive, and accessible care, leveraging digital health tools such as mobile apps may help fill the gap in addressing the unique spiritual needs of YAs with cancer and provide opportunities for efficacious, scalable interventions to increase access and reach to YAs who are most in need. Currently, research on interventions (digital or otherwise) to support spiritual wellbeing in YAs with cancer is exceedingly rare. This feasibility work will be a first step in testing whether a spiritual self-care mobile app can be used to support spiritual wellbeing in YAs with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Young adults between the ages of 18 and 39
* Histologically confirmed diagnosis of cancer (except basal cell skin carcinoma)
* For patients with solid tumors, patients must be within 12-weeks of current cancer diagnosis upon enrollment and currently receiving curative treatment (i.e., surgery and/or chemotherapy and/or radiation therapy; surgery-only patients must be within 6-weeks of surgery at time of enrollment). For patients with hematological cancers, there is no requirement for time since diagnosis, provided they are receiving treatment, including stable maintenance management.
* Able to provide informed consent and fluent in English for completion of study questionnaires
* Residing in the USA
* Internet access
* Own a smartphone with an active data plan or wi-fi
* Have a personal email address

Exclusion Criteria:

* Unable to provide informed consent
* Not currently engaging in curative cancer treatment(s) (i.e., awaiting treatment initiation, completed curative treatment(s))
* Currently receiving end-of-life palliative care or hospice care

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Acceptability of spiritual self-care smartphone app | Week 6
  At the end of each week of the 6-week intervention, participants will complete a brief survey to self-report: a) acceptability of the app (i.e., how enjoyable, beneficial, difficult, were your interactions with the content measured on scale of 0%-not at all to 100%-very much), b) preferred time of day, c) preferred content, d) intentions to continue use, and e) barriers and facilitators to use during the past week. At the end of the intervention period, we will assess overall acceptability of the app (i.e., how enjoyable, beneficial, difficult, etc. was the intervention overall measured on scale of 0%-not at all to 100%-very much; how likely are you to recommend this to a friend/someone with cancer).
Demand of spiritual self-care smartphone app | Week 10
  Study accrual and retention rates (i.e., number of participants screened, enrolled, and withdrawn throughout the study) and user statistics of app use during the 6-week study period (i.e., total number of minutes of app use per day, count of sessions per day, total days of app use).

SECONDARY OUTCOMES:
Expectancy ratings of spiritual self-care smartphone app | Baseline
  Baseline expectancy before engaging with the app (i.e., how enjoyable, beneficial, difficult, do you think this intervention will be? measured on a scale of 0%-not at all to 100%-very much - higher score denoting higher acceptance) and confidence in intentions to use the app daily.
Spiritual Wellbeing Scores | Baseline, Week 6, and Week 10 (follow-up)
  12-item Functional Assessment of Cancer Therapy - Spiritual Wellbeing (FACIT-Sp-12). Includes 12 items scored on a scale of 0 (not at all) to 4 (very much). A total score and 3 subscale scores (i.e., faith, meaning, peace) can be calculated with higher scores indicating greater levels of spiritual wellbeing (Scores range from 0-36)
Life Satisfaction Scores | Baseline, Week 6, and Week 10 (follow-up)
  NIH Toolbox short form assessing life satisfaction. 5 items scored on a scale of 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater life satisfaction (Scores range from 5-35)
Positive Affect Scores | Baseline, Week 6, and Week 10 (follow-up)
  NIH Toolbox short form assessing positive affect. 15 items scored on a scale of 1 (not at all) to 5 (very much). Higher scores indicate greater positive affect.
Self-Efficacy Scores | Baseline, Week 6, and Week 10 (follow-up)
  PROMIS short form assessing general self-efficacy. 4 items scored on a scale of 1 (I am not at all confident) to 5 (I am very confident). Higher scores indicative of higher levels of self-efficacy.
Health-Related Quality of Life Scores | Baseline, Week 6, and Week 10 (follow-up)
  PROMIS AYA Health Status Profile to capture health-related quality of life domains, including depression, anxiety, fatigue, physical function, pain interference, emotional support, and cognitive function, and pain intensity.
Qualitative Interviews | Week 6
  A subsample of participants (~10-12) will be asked to discuss their attitudes about the app, internal and external factors that prevented them from using the app when they intended to, along with the factors that supported their use of the app.

CONTACTS AND LOCATIONS:
Overall Officials: John M Salsman, PhD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No
Pilot data that is descriptive in nature